CLINICAL TRIAL: NCT06780371
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Kinesiophobia and Pressure Sore Risk After Bariatric Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Okutan3
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Kinesiophobia; Pressure Sore; Emotional Freedom Technique; Complementary Therapies; Bariatric Surgery
Keywords: pressure sore; Kinesiophobia; emotional freedom technique
MeSH Terms: conditions — Kinesiophobia; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-test-post-test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): After the pre-test application (Personal Introduction Form, Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) EFT was applied to the patients when they were stable before the bariatric surgery and they were taught to do it on their own. After the bariatric surgery, the patients were asked to do 1 session of EFT and were accompanied. After the application, the patients were applied post-tests (Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale). EFT training was given by a researcher who has a certificate in the field.
  Interventions: Other: Emotional Freedom Technique
- No Intervention: Control Group (No Intervention): Pre-tests were administered to patients (Personal Introduction Form, Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) at a stable time before bariatric surgery. Post-tests (Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) were administered to patients (Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) at a stable time after bariatric surgery. After the post-tests, EFT was administered to patients in the control group.

INTERVENTIONS:
Other: Emotional Freedom Technique — Emotional Freedom Technique application; It is an application that works on cognitive and energetic levels.
  Emotional Freedom Technique Application Instructions
  1. Determination of Subjective Units of Disturbance (SUD)
  2. Preparation or setup
  3. Application of appropriate acupuncture points in order
  4. 9-Gamut: An application that allows the two hemispheres of the brain to be stimulated simultaneously
  5. Application of appropriate acupuncture points in order again
  6. Control of the differentiation in the level of discomfort with SUDS again
  Arms: Experimental: Intervention Group

SUMMARY:
The aim of this study was to investigate the effect of emotional freedom technique on kinesiophobia and the risk of developing pressure sores in patients undergoing obesity surgery.

The hypotheses of the study are as follows:

H1-0: Emotional liberation technique has no effect on kinesiophobia in patients undergoing bariatric surgery.

H1-1: Emotional liberation technique has a positive effect on kinesiophobia in patients undergoing bariatric surgery.

H2-0: Emotional liberation technique has no effect on the risk of developing pressure ulcers in patients undergoing bariatric surgery.

H2-1: Emotional liberation technique has a positive effect on the risk of developing pressure ulcers in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Intervention Group: After the pre-test application (Personal Introduction Form, Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) EFT was applied to the patients when they were stable before the bariatric surgery and they were taught to do it on their own. After the bariatric surgery, the patients were asked to do 1 session of EFT and were accompanied. After the application, the patients were applied post-tests (Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale). EFT training was given by a researcher who has a certificate in the field.

Control Group Patients were administered pre-tests (Personal Introduction Form, Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) at a stable time before bariatric surgery. Post-tests (Tampa Kinesiophobia Scale and Braden Pressure Sore Risk Assessment Scale) were administered to patients after bariatric surgery at a stable time. After the post-tests, EFT was administered to patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older
2. Having had obesity surgery
3. Not having any visual or auditory problems
4. Not having any psychiatric problems.

Exclusion Criteria:

1. Not accepting to participate in the study or wanting to leave
2. Being under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
kinesiophobia level | 20 minutes
  It is a scale that measures movement restriction. As a result of the survey, the person receives a total score between 17-68 according to the answers they give. A high score on the scale indicates that the person has a high level of kinesiophobia. Those with a score above 37 are grouped as "high level kinesiophobia", those with a score of 37 and below are grouped as "low level kinesiophobia"
pressure ulcer risk | 20 minutes
  The Braden Scale was developed in 1987 by Nancy Bergstrom, Barbara J. Braden and their colleagues for the early diagnosis of patients at risk of pressure ulcers.
  The lowest score that can be obtained from the scale is 6, and the highest score is 23. Patients who receive 12 points or less from the scale are considered high risk, 13-14 points are considered risky, 15-16 points are considered low risk, and 15-18 points are considered low risk in patients over the age of 75

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, PhD., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)